CLINICAL TRIAL: NCT01897402
Title: A Phase 2 Double Blind Study to Evaluate Safety and Immunogenicity of Meningococcal Meningitis Serogroups A, C, Y & W-135 Polysaccharide Diphtheria Toxoid Conjugate Vaccine (NmVac4-A/C/Y/W-135-DT™) Compared With a Licensed Vaccine
Brief Title: Immunogenicity and Safety of Group A, C, Y & W-135 Meningococcal Polysaccharide Diphtheria Toxoid Conjugate Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JN-International Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JN-NM-002
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Meningococcal Meningitis; Meningococcal Infections
Keywords: Central Nervous System Infections; Meningitis; toxoid; Meningococcal vaccine; conjugate vaccines
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections; Central Nervous System Infections; Meningitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Vaccine (Experimental): NmVac4-A/C/Y/W-135-DT™ conjugate vaccine
  Interventions: Biological: Test Vaccine
- US Licensed Vaccine (Active Comparator): Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine
  Interventions: Biological: US Licensed Vaccine

INTERVENTIONS:
Biological: Test Vaccine — NmVac4-A/C/Y/W-135-DT™ conjugate is a vaccine in liquid form composed of purified polysaccharides (PS) conjugated to diphtheria toxoid. Single intramuscular 0.5 mL dose contains 4 µg each of Serogroup A, C, W-135, and Y PS conjugated to approximately 26 µg total diphtheria toxoid.
  Other Names: meningococcal meningitis conjugate vaccine, quadrivalent; NmVac4-A/C/Y/W-135-DT™
  Arms: Test Vaccine
Biological: US Licensed Vaccine — Meningococcal (Groups A,C,Y,W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine 0.5 mL dose, intramuscular. Single dose contains 4 µg each Serogroup A, C, W-135 and Y conjugated to approximately 48 µg total diphtheria toxoid.
  Other Names: meningococcal meningitis conjugate vaccine, quadrivalent
  Arms: US Licensed Vaccine

SUMMARY:
The purpose of this study is to evaluate the production of antibodies to a new conjugate vaccine, NmVac4-A/C/Y/W-135-DT, as a measure of vaccine effectiveness, compared to the production of antibodies to a similar, licensed meningococcal (Groups A, C, Y, W-135) polysaccharide diphtheria toxoid (DT) conjugate vaccine. The investigators will also evaluate the safety of NmVac4-A/C/Y/W-135-DT™ conjugate vaccine compared to the licensed vaccine. The hypothesis is that the test vaccine is comparable to the licensed active control vaccine.

DETAILED DESCRIPTION:
Meningococcal disease is a potentially life-threatening bacterial infection. The disease most commonly is expressed as either meningococcal meningitis, an inflammation of the membranes surrounding the brain and spinal cord, or meningococcemia, the presence of bacteria in the blood. The most common symptoms include high fever, headache, neck stiffness, confusion, nausea, vomiting, lethargy, and rash. If not treated the disease can progress rapidly and can lead to shock and death, often within hours of the onset of symptoms. The disease is fatal at a rate of 10%. Of patients who recover, 10% have permanent hearing loss or other serious sequelae.

Neisseria meningitidis capsular polysaccharides are poor immunogens. However, conjugation of bacterial polysaccharides to immunogenic carrier proteins generally results in conjugates that induce strong anti-polysaccharide T-helper cell dependent immune responses, creating a longer-lasting immune response and thus protection against meningococcal infection.

The sponsor's small size Phase 1 clinical trial comprised 60 subjects. Therefore, additional data is needed to confirm the previous data with a statistically powered Phase 2 clinical trial. The present study aims to evaluate subject responses to single doses, administered in adult subjects, to determine further safety and immunogenicity of the vaccine. This study compares safety and antibody production induced by one intramuscular injection of either NmVac4-A/C/Y/W-135-DT or a licensed meningococcal (Groups A, C, Y, W-135) polysaccharide diphtheria toxoid conjugate vaccine. The primary immunogenicity endpoint will be seroresponse, based on antibody titer ≥1:8 for subjects with titer <1:8 at baseline or a 4-fold rise in antibody levels, 4 weeks after a single injection . The number and proportion of subjects achieving seroresponse will be tabulated by serogroup for each vaccine group. A non-inferiority test will be used to determine if the immune response elicited by NmVac4 A/C/Y/W-135-DT™ is not less than a specified difference in percent seroconversion from the licensed control vaccine. Participants will attend a screening visit up to 6 weeks prior to vaccination (day 0), then will attend study visits for 4 weeks. There will be a study phone call at days 2-3, then a post-study call to subjects to assess safety at 26 weeks.

ELIGIBILITY:
Inclusion Criteria (IC):

* Participant is willing and able to give informed consent and comply with all aspects of the evaluation after the nature of the study is explained.
* Male or female, aged 18 to 55 years old
* In general good health with no significant chronic or acute conditions that would interfere with immune response or expected Adverse Event (AE) evaluation in the opinion of the investigator as determined by Medical history and/or History-directed physical examination
* Abstinence or use of effective contraception by the participants or their partners during the trial and continuing for four weeks after vaccination will be required for males or female participants of child bearing potential.
* Able (in the opinion of the investigator) to comply with all study requirements.

Exclusion Criteria (EC):

* Unwilling or unable to understand study requirements and give written informed consent for the study.
* Prisoners.
* History of Guillain-Barré syndrome (GBS).
* Pregnancy (confirmed by positive pregnancy test) or lactation.
* Previous diagnosis of laboratory confirmed meningococcal disease.
* Previous meningococcal meningitis vaccination in the last five years
* Laboratory abnormalities that are considered Grade 2 or higher (based on AE, ranges as described in the protocol appendix) that in the opinion of the Investigator would raise safety concerns for participation in the study or interfere with evaluation of study objectives, or abnormalities >2 times the Upper Limit of Normal range (ULN).
* Known or suspected autoimmune or connective tissue disorders, including rheumatoid arthritis and congenital or acquired immunodeficiency. Does not include mild to moderate seasonal/perennial allergies treated with over the counter antihistamines.
* Use of systemic immunosuppressive drugs or therapy within 6 months prior to study enrollment, not including topical or inhaled steroids/cytotoxic agents. Includes anti-cancer chemotherapy, radiation, and long term systemic corticosteroid therapy. History of anaphylactic shock, severe asthma, urticaria, or other allergic or hypersensitivity reactions following vaccination or known hypersensitivity to any vaccine component.
* Received blood, blood products, plasma derivatives or any parenteral immunoglobulin preparation in the past 3 months.
* Use of systemic antibiotics within 72 hours prior to study enrollment.
* History of cirrhosis or hepatitis.
* Known bleeding disorder or condition associated with a prolonged bleeding time.
* Positive results of testing for hepatitis B surface antigen (HepBsAg), Hepatitis C or HIV-1 or HIV-2 antibodies. Known or suspected HIV or Hepatitis B or C infection.
* Positive results of drug screen that cannot be explained by use of approved prescription medication (amphetamine, tetrahydrocannabinol (THC), cocaine). Current (past 30 days) heavy smokers (greater than or equal 1 pack per day).tetrahydrocannabinol
* Received another investigational product within the last 30 days. Investigational product may be a drug, vaccine, medical device or medical procedure.
* History of significant head trauma, alcohol or substance abuse or other medical illnesses that could cause a neurological deficit (e.g., cerebro-vascular disease).
* Medication or alcohol use that, in the opinion of the Investigator, may influence or bias the clinical outcome of the trial.
* History of any serious chronic medical or psychiatric illnesses or condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.
* History of chronic or severe headaches, myalgia, arthralgia, malaise, fatigue or other systemic disorder commonly observed as AEs for licensed meningococcal vaccines.
* Currently experiencing a cold, flu or other acute illness (subject may be deferred until after recovery).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 525 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Yataco, MD, Principal Investigator — IRC Clinics,; Jeffrey E Atkinson, MD, Principal Investigator — Chesapeake Research Group; Myron I Murdock, MD, Principal Investigator — Mid Atlantic Urology Associates LLC
Locations (3):
- United States (3):
  - Mid Atlantic Urology Associates LLC, Greenbelt, Maryland
  - Chesapeake Research Group, Pasadena, Maryland
  - IRC Clinics, Towson, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited and were enrolled at three sites in Maryland between October 21, 2013 and May 22, 2014. The sites screened 1086 subjects with 559 screen failures. The majority, 390 subjects (69.8 %), failed due to inclusion or exclusion criteria (IC/EC). The most common failure criterion was Laboratory abnormalities (150 subjects, 26.8 %).
Pre-assignment Details: Other common reasons for screen failure were inability to re-schedule within enrollment window after trial start was delayed (101 subjects, 18.1 % of screen failures) and lost to follow up 65 subjects (11.6%). These two reasons account for 166 (29.7%) subjects who met IC/EC, but did not enter the trial.
Period: Overall Study
Arm/Group | Test Vaccine | US Licensed Vaccine
Started | 265 | 260
Completed | 246 | 244
Not Completed | 19 | 16

BASELINE CHARACTERISTICS:
Population: Population contains all randomized subjects. Two randomized subjects could not be vaccinated. Three subjects, one female and 3 males received incorrect vaccine. They are listed according to randomized treatment in the baseline population, but were analyzed according to the actual vaccine received in the safety population (secondary outcomes).
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Vaccine | US Licensed Vaccine | Total
Number analyzed (Participants) | 266 | 261 | 527
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (11.1) | 36.0 (10.88) | 36.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 112 | 228
  Male | 150 | 149 | 299
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 3 | 4
  American Indian/ Alaska Native | 0 | 2 | 2
  Caucasian | 87 | 89 | 176
  Black/ African-American | 176 | 160 | 336
  Native Hawaiian/Pacific Islander | 0 | 0 | 0
  Hispanic or Latino | 2 | 6 | 8
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Seroresponse (Percent Seroconversion).
Description: Rise in antibody titers in serum at 4 weeks after vaccination, compared to baseline titer for meningococcal serogroups A, C, Y, and W-135. Serum Bactericidal Assay with human complement: Antibody titer ≥1:8 for subjects with titer <1:8 at baseline or a 4-fold rise in antibody levels.
Time Frame: Week 4 after injection
Population: Per Protocol Population
Measure: Number (95% Confidence Interval); unit: percentage of per protocol participants
Arm/Group | Test Vaccine | US Licensed Vaccine
Number analyzed (Participants) | 222 | 226
percentage of per protocol participants
  Serogroup A | 70.7 [64.3 to 76.6] | 70.1 [63.6 to 76.1]
  Serogroup C | 66.5 [59.9 to 72.7] | 72.5 [66.1 to 78.3]
  Serogroup Y | 63.1 [56.3 to 69.4] | 64.1 [57.5 to 70.4]
  Serogroup W-135 | 66.2 [59.6 to 72.4] | 65.9 [59.3 to 72.1]
Statistical Analysis 1: Comparison: Test Vaccine vs US Licensed Vaccine; The hypothesis was that the test vaccine is comparable to the licensed active control vaccine. Differences between treatment groups were described using exact two-sided 95% confidence intervals on differences in % seroconversion between the two treatment groups (test vaccine minus reference vaccine) for each serogroup. If the lower bound of the difference is ≥ -15%, then the test vaccine meets the preliminary criterion for non-inferiority; Test type: Non-Inferiority or Equivalence — The assumptions for the sample size calculations were: 1) Seroconversion for the control vaccine (Menactra) is 40-80% and 2) the true treatments are theoretically equal and 3) the power of detecting non-inferiority is 90%; Percentage Difference = 0.6, 95% CI 2-sided [-7.9 to 9.1] — Serogroup A
Statistical Analysis 2: Comparison: Test Vaccine vs US Licensed Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Percentage Difference = -6.0, 95% CI 2-sided [-14.6 to 2.6] — Serogroup C
Statistical Analysis 3: Comparison: Test Vaccine vs US Licensed Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Percentage Difference = -1.0, 95% CI 2-sided [-9.9 to 7.9] — Serogroup Y
Statistical Analysis 4: Comparison: Test Vaccine vs US Licensed Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Percentage Difference = 0.3, 95% CI 2-sided [-8.5 to 9.1] — Serogroup W-135

2. Secondary Outcome: Solicited Adverse Events From Diary Cards
Description: Local and systemic rates from Diary Cards filled by the participants.
Time Frame: Day 0 to Day 7 after vaccination
Population: Safety Population: All vaccinated participants, grouped by actual vaccine received.
Measure: Number; unit: percentage of participants
Groups:
- Test Vaccine - Male; Test Vaccine - Female: NmVac4-A/C/Y/W-135-DT™ conjugate vaccine
- US Licensed Vaccine - Male; US Licensed Vaccine - Female: Meningococcal (Groups A, C, Y and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine
Arm/Group | Test Vaccine - Male | Test Vaccine - Female | US Licensed Vaccine - Male | US Licensed Vaccine - Female
Number analyzed (Participants) | 151 | 114 | 147 | 113
percentage of participants
  At least 1 local reaction | 53.6 | 65.8 | 40.8 | 46.5
  At least 1 systemic reaction | 35.1 | 37.7 | 34.7 | 42.5

3. Secondary Outcome: Non Solicited Adverse Events
Description: Non solicited local and systemic adverse Event (AE) rates throughout the course of the study, based on laboratory test results, vital signs, examination and questioning the subjects.
Time Frame: up to 6 months
Population: Safety Population: All vaccinated participants, grouped by actual vaccine received.
Measure: Number; unit: participants
Arm/Group | Test Vaccine | US Licensed Vaccine
Number analyzed (Participants) | 265 | 260
participants
  Subjects with at least 1 AE | 45 | 54
  Subjects with at least 1 treatment related AE | 1 | 5

ADVERSE EVENTS:
Time Frame: Solicited AEs: vaccination day and 7 days following vaccination (participant diary cards, Outcome 2). AEs were also collected at each visit (4 weeks) and by phone calls 2-3 day following vaccination and at 6 months following vaccination (Outcome 3).
Description: Methods: standard questionnaire, investigator assessment, laboratory testing, scheduled telephone calls.
  Solicited AEs (secondary outcome 2) and non solicited AEs (secondary outcome 3) are included in the other adverse event totals. All AEs meeting the 4% threshold except increased blood pressure were solicited AEs from diary cards.
Arm/Group | Test Vaccine | US Licensed Vaccine
Serious Adverse Events (participants affected / at risk) | 0/265 | 1/260
Other Adverse Events (participants affected / at risk) | 173/265 | 141/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Vaccine (N=265) | US Licensed Vaccine (N=260)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) — Not associated with the vaccine. All 3 Serious Adverse Events affected the same subject.
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) — Not associated with the vaccine. All 3 Serious Adverse Events affected the same subject.
Glomerular Filtration Rate Decreased (Investigations) | 0 (0) | 1 (1) — Not associated with the vaccine. All 3 Serious Adverse Events affected the same subject.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Vaccine (N=265) | US Licensed Vaccine (N=260)
Tenderness around injection site (General disorders) | 134 | 100 — Local from Dairy Cards
Pain around injection site (General disorders) | 109 | 86 — Local from Dairy Cards
Myalgia (Musculoskeletal and connective tissue disorders) | 53 | 49 — Systemic from Dairy Cards
Headache (Nervous system disorders) | 46 | 40 — Systemic from Dairy Cards
Fatigue (General disorders) | 43 | 42 — Systemic from Dairy Cards
Hardness around injection site (General disorders) | 37 | 26 — Local from Dairy Cards
Swelling around injection site (General disorders) | 35 | 23 — Local from Dairy Cards
Malaise (General disorders) | 24 | 26 — Systemic from Dairy Cards
Diarrhea (Gastrointestinal disorders) | 22 | 20 — Systemic from Dairy Cards
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 21 — Systemic from Dairy Cards
Nausea (Gastrointestinal disorders) | 25 | 15 — Systemic from Dairy Cards
Chills (General disorders) | 19 | 14 — Systemic from Dairy Cards
Anorexia (Metabolism and nutrition disorders) | 18 | 12 — Systemic from Dairy Cards
Blood Pressure Systolic Increased (Investigations) | 16 | 12 — Systemic

LIMITATIONS AND CAVEATS:
Three subjects, 1 female and 2 males, received incorrect vaccine. They are listed according to randomized treatment in the baseline population, but were analyzed according to the actual vaccine received in the safety population (outcomes 2 and 3).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All abstracts, presentations or manuscripts, and any data analyses conducted independently by the Investigator must be submitted in advance to the sponsor for review and approval. The sponsor will not unreasonably withhold publication of study findings. The objective of this policy is to ensure consistency between data filed with a regulatory authority and those appearing in the publication.